CLINICAL TRIAL: NCT05549193
Title: The Effects of the Pelvic Floor and Abdominal Muscle Training in Urinary Incontinence According to the Severity
Brief Title: The Effects of the Pelvic Floor and Abdominal Muscle Training on Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ilke Keser, Principal Investigator, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24074710-604.01.01-44
Record Dates: First submitted 2022-09-12; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Urinary Incontinence
Keywords: Rectus Abdominus; Pelvic Floor Muscle Training; Stress Urinary Incontinence; Quality of Life; Biofeedback; Home Exercises
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild and Moderate-Severe Urinary Incontinence Group (Experimental): 10 sets of pelvic floor muscle training and 2 sets of abdominal muscle strengthening training were given every day for 6 weeks. All analyzes were conducted at the beginning and end of the 6-week training. The same training program was applied to both groups ( Group 1 (mild urinary incontinence) and Group 2 (moderate-severe urinary incontinence), and the effects were compared according to the severity of incontinence.
  Interventions: Other: Exercises Training

INTERVENTIONS:
Other: Exercises Training — Pelvic Floor Muscle Training: For slow contractions, it was asked to contract in 5 seconds gradually, wait at a maximum of 5 seconds and gradually relax in 5 seconds. For fast contractions, it was asked to contract at a maximum of 2 seconds and then to relax. 10 fast + 10 slow contractions were accepted as 1 set exercise. (10 sets x Every Day x 6 weeks)
  Transversus Abdominus: Patients were in the crook lying position and were asked to contract their abdominal muscles strongly and statically. 15 repetitions were carried out, each consisting of contraction for 10 s and relaxation for 20 s. 2 sets of 15 repetitions were done.
  Internal Obliquus Abdominus: Patients were in the crook lying position and were asked to contract their abdominal muscles strongly and statically and then try to touch the furthest point of their legs with their fingertips for 15 repetitions consisting of contraction for 10 s followed by relaxation for 20 s. The sequence was then repeated on the other leg.

SUMMARY:
To investigate the effects of the pelvic floor and abdominal muscle training on the severity of incontinence in women with stress and mixed urinary incontinence.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of incontinence severity on the pelvic floor and abdominal muscle strengthening training in women with stress urinary incontinence (UI). Sixteen patients with stress and mixed UI were included in the study. According to the 24-hour pad test (24hPT), individuals were divided into two groups as group 1 (24hPT 4-20gr, mild group, n: 9) and group 2 (24hPT 21g and above in 24hPT, moderate-severe group, n: 7). Pelvic floor muscle training (PFMT) and abdominal muscle training were applied to the groups for 6 weeks.

PFMT was given as a home-based exercise program to increase pelvic floor muscle (PFM) strength and endurance. Before starting the program, PFM was taught first schematically and then by the biofeedback method. It was ensured that the patient learned the PFM. Fast and slow pelvic floor contractions were taught for both type 1 and type 2 muscle fibres. For slow contractions, it was asked to gradually contract in 5 seconds, wait at a maximum of 5 seconds and gradually relax in 5 seconds. For fast contractions, it was asked to contract at a maximum of 2 seconds and then to relax. Patients were asked to perform 10 slow contractions after every 10 rapid contractions. 10 fast + 10 slow contractions were accepted as 1 set exercise. Subjects were asked to make 10 sets every day for 6 weeks.

Strengthening exercises for transversus abdominus and internal obliques abdominus muscles were given as a home program and the details were written below:

Transversus Abdominus: Patients were in the crook lying position and were asked to contract their abdominal muscles strongly and statically. Fifteen repetitions were carried out; each one consisting of contraction for 10 s followed by relaxation for 20 s. After 15 repetitions, patients rested for 5 min. The sequence was then repeated for two sets of 15 repetitions.

Internal Obliquus Abdominus: Patients were in the crook lying position and were asked to contract their abdominal muscles strongly and statically and then try to touch the furthest point of their legs with their fingertips for 15 repetitions consisting of contraction for 10 s followed by relaxation for 20 s. After 15 repetitions, patients rested for 5 min. The sequence was then repeated on the other leg.

Urinary incontinence, pelvic floor muscle strength measurement, quality of life, symptom, and the presence of pelvic floor dysfunction were evaluated respectively using 24hPT, Electromyography (EMG) Biofeedback device, King's Health Questionnaire, Urogenital Distress Inventory, and Global Pelvic Floor Bother Questionnaire. Evaluations were performed at the beginning and at the end of the physiotherapy program, and a subjective improvement rate was determined.

ELIGIBILITY:
Inclusion Criteria:

* Being female,
* Being 18 years of age or older
* Having been diagnosed of SUI and stress-predominant MUI after urodynamic evaluation by the urologist.

Exclusion Criteria:

* Currently taking medications for UI,
* Having urinary tract infection,
* Neurological disorders,
* Pelvic organ prolapse stage >2,
* Pregnancy,
* a mental problem and/or
* been applied prior to physiotherapy for UI.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with incontinence diagnoses were referred by the doctor. Gender identity is based on patients' self-representation and anatomical structures.
Enrollment: 16 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence Severity | 6 weeks
  A 24-hour pad test was used to assess and standardize the severity of UI. The patients were informed before the test. The patients were told to change their pads every 4-6 hours and put the pads in an airtight locked bag to prevent the urine from evaporating. Since the pads should be weighed immediately after the evaluation, they were asked to do the test 1 day before the evaluation. Pads that were used for 24 hours were requested in a mouth-locked bag. 1 unused pad of the same type was requested. Urinary incontinence was determined by measuring the weight of the pad with precision scales (Isolab Laborgerate GMBH, Germany) before and after 24 hours. As a result of the 24-hour pad test, 4-20 grams were defined as mild, 21-74 grams as moderate, and > 75 grams as severe UI.

SECONDARY OUTCOMES:
Pelvic Floor Muscle Activity | 6 weeks
  Muscle activity in electromyography was evaluated by the EMG Biofeedback program of MMS brand Uro Solar Model urodynamics device (Medical Measurement Systems b.v. the Netherlands). Superficial electrodes were used for the measurement. Electrodes were non-invasively measured by adhering 2 pieces to the right and left of the perineal body and 1 to the inner leg. EMG values were recorded. Evaluations were made with the patient in the lithotomy position. During the measurement, it was warned that the PFM should contract for 10 seconds and during contractions they should not contract the abdominal, hip and thigh muscles and hold their breath. For correct contraction, patients were asked to breathe normally and then to squeeze and lift the pelvic floor as if preventing the escape of urine or flatus. Muscle activation response recorded in microvolts (μV).
Abdominal Muscles Strength | 6 weeks
  To assess abdominal muscle strength, Dr Robert W. Lovett's manual muscle test was used. It was started with the value 3, and patients that can make the value of 3 were examined with 3+, 4, and 5 values of the muscle. If the patients cannot make 3, 2, 1, and 0 values were examined. All tests were performed by the same physiotherapist according to a standardised protocol.
Quality of life about Urinary Incontinence | 6 weeks
  King's Health Questionnaire was used to assess the quality of life specific to UI. It consists of two parts and 32 items.
Urinary Incontinence Symptom severity | 6 weeks
  The Urinary Distress Inventory-short form was used to evaluate the symptom severity score. It consisted of 6 questions and each question was scored between 0-3 points. If the scoring is high, the quality of life is low.
Existing pelvic floor dysfunction | 6 weeks
  Global Pelvic Floor Bother Questionnaire was used to determine how much pelvic floor dysfunction exists. The questionnaire consists of 9 questions and if the scoring is high, the complaint is high.
Treatment adherence | 6 weeks
  At the beginning of the treatment, an exercise follow-up form was given, and the patients were asked to mark it regularly. In the final evaluation, follow-up forms were obtained from the patients. During the treatment, the patients were followed up every week by phone. The compliance and continuity of the patients were followed closely. Patients who missed more than 2 treatments were excluded from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)